CLINICAL TRIAL: NCT07388810
Title: Study of Different Doses of Ripertamab in Children With Frequent Relapses or Steroid-Dependent Nephrotic Syndrome：An Open-label Randomized Controlled Trial
Brief Title: Study of Ripertamab in Children With Frequent Relapses or Steroid-Dependent Nephrotic Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mao Jianhua (Other)
Collaborators: Sinocelltech Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Mao Jianhua, Professor, The Children's Hospital of Zhejiang University School of Medicine
Organization: The Children's Hospital of Zhejiang University School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCT400-NS-ch
Record Dates: First submitted 2026-01-29; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: FRNS/SDNS; Ripertamab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Two doses group (Experimental): 2 doses of 375mg/m2 BSA ripertamab at 1-week intervals( within ±1days).
  Interventions: Drug: ripertamab
- One dose group (Active Comparator): 1 dose of 375mg/m2 BSA ripertamab.
  Interventions: Drug: ripertamab

INTERVENTIONS:
Drug: ripertamab — 2 doses of 375mg/m2 BSA ripertamab at 1-week intervals( within ±1days). At the meantime, prednisone is administered at a dose of 1.5 mg/kg/d (maximum 40 mg) on alternate days or at the dose being used every alternate day before randomization. After 2 weeks, the dose is reduced by 0.25 mg/kg every 2 weeks, and the drug is discontinued at 3 months.
  Arms: Two doses group
Drug: ripertamab — 1 dose of 375mg/m2 BSA ripertamab. At the meantime, prednisone is administered at a dose of 1.5 mg/kg/d (maximum 40 mg) on alternate days or at the dose being used every alternate day before randomization. After 2 weeks, the dose is reduced by 0.25 mg/kg every 2 weeks, and the drug is discontinued at 3 months.
  Arms: One dose group

SUMMARY:
This is an open-label randomized controlled trial to evaluate the efficacy and safety of one dose versus two doses of ripertamab in children with frequent relapses or steroid-dependent nephrotic syndrome (FRNS/SDNS).

ELIGIBILITY:
Inclusion Criteria:

1. 16 years old and above with FRNS/SDNS
2. Before enrollment, achieved complete remission (urine protein/creatinine ratio (morning urine or 24-hour urine) ≤ 20mg/mmol (0.2mg/mg) or < 100mg/m2/d, or test strip result negative or trace)
3. Within 2 months before enrollment, did not use levamisole, alkylating agents such as cyclophosphamide, calcineurin inhibitors such as cyclophosphamide and cyclosporine, or mycophenolate mofetil. Within 6 months before enrollment, did not use other CD20 monoclonal antibodies (such as ofatumumab, otuzumab, etc., excluding rituximab)
4. Glomerular filtration rate (eGFR) > 60ml/min/1.73m2
5. The patient or their guardian agrees to participate in this clinical trial and signs the informed consent form, indicating that they understand the purpose and procedures of this clinical trial and are willing to participate in the study

Exclusion Criteria:

1. Known causes (such as systemic lupus erythematosus, IgA nephropathy, other secondary nephrotic syndromes, amyloidosis, malignant tumors, etc.)
2. Known active chronic infections, including tuberculosis, HIV, HBV, HCV, etc.
3. Severe leukopenia (white blood cells < 3.0×109/L), severe anemia (hemoglobin < 8.9 g/dl), thrombocytopenia (platelets < 100×109/L), or liver dysfunction (alanine aminotransferase/aspartate aminotransferase > 2 times the upper limit of normal)
4. Received live vaccines within 1 month prior to screening
5. Currently participating in other drug clinical trials
6. Other conditions that the investigator deems make the patient unsuitable for this study

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 312 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Relapse free survival rate | 1 year
  Relapse free survival rate at 1 year

SECONDARY OUTCOMES:
Recurrence frequency at 6 and 12 months | 1 year
  Recurrence frequency within 6 months during the study period. Recurrence frequency within 12 months during the study period.
Cumulative corticosteroid dose | 1 year
  Total amount of corticosteroids used in 1 year during the study period
Median recurrence-free survival | 18 months
  From admission day to 18 months
B-cell count | 18 months
The occurrence and severity of adverse events | 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang Province 310052, Hangzhou, Zhejiang, China